CLINICAL TRIAL: NCT00394940
Title: Serum Inflammatory Biomarkers as Predictors of COPD Morbidity and Mortality
Brief Title: Identifying Inflammatory Biomarkers of Chronic Obstructive Pulmonary Disease
Status: Completed | Type: Observational
Sponsor: University of Arizona (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Stefano Guerra, Associate Research Professor, University of Arizona
Other Study IDs: 1349; R21HL085195-01 (NIH)
Record Dates: First submitted 2006-10-31; First posted 2006-11-02 (Estimated); Last update posted 2017-12-06 (Actual); Status verified 2017-12

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Emphysema; Chronic Bronchitis; Inflammation; CD14; TLR4; Proteomics
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema; Bronchitis, Chronic; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA, serum, supernatants
Oversight: Data Monitoring Committee: No

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a condition that is characterized by airway obstruction due to inflammation. Levels of inflammatory proteins may be linked to when and to what extent COPD develops. This study will use data collected during the Tucson Epidemiological Study of Airway Obstructive Disease (TESAOD) and its 33-year follow-up to determine the relationship between inflammatory protein expression and COPD.

DETAILED DESCRIPTION:
COPD is a term that encompasses both chronic bronchitis and emphysema, two diseases that are characterized by airway obstruction that interferes with normal breathing. Airway inflammation can stem from exposure to harmful fumes in the air, chronic bacterial infections in the airways, and a genetic predisposition to an inflammatory response to these agents. In people with COPD, the airway inflammation may extend beyond the lungs and contribute to systemic symptoms and, ultimately, to an increased mortality risk. Markers of systemic inflammation have been identified, but the relationship between these markers and when and to what extent COPD develops has not been determined. This study will use data collected during the TESAOD and its 33-year follow-up to determine the relationship between COPD and the expression of various inflammatory proteins, including pro-inflammatory cytokines (e.g., IL-6, IL-8, TNF-alpha) and acute phase proteins (e.g., C-reactive protein, soluble CD14).

This study will not recruit any new participants. Detailed respiratory phenotypic information and serum samples that were collected during the TESAOD study will be evaluated in conjunction with newly generated biomarker and protein information. No new phenotypic data or biological specimens will be collected in this study.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in the Tucson Epidemiological Study of Airway Obstructive Disease (TESAOD)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Sample of the general population that was enrolled in 1972
Sampling Method: Probability Sample
Enrollment: 2085 (Actual)
Dates: Start 2006-07; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
COPD development defined as FEV1/FVC < 70% | up to 50 years

SECONDARY OUTCOMES:
COPD progression defined based on decline of lung function | up to 50 years
Mortality | up to 50 years

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Guerra, MD, PhD, Principal Investigator — Arizona Respiratory Center
Locations (1):
- Arizona Respiratory Center, Tucson, Arizona, United States

REFERENCES:
- See also: Click here for the Arizona Respiratory Center Web site — http://www.arc.arizona.edu/